CLINICAL TRIAL: NCT04417738
Title: Unilateral Transcranial Photobiomodulation for the Treatment of Opioid Cravings: A Blinded Placebo-Controlled Evaluation of Efficacy and Safety
Brief Title: Transcranial Photobiomodulation for the Treatment of Opioid Cravings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MindLight, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NEIRB001
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2020-06

CONDITIONS: Opioid-use Disorder; Depression, Anxiety; Craving
Keywords: opioid craving; opioid use disorder; depression; anxiety; transcranial photobiomodulation; near infra-red light; dual-brain psychology; cerebral laterality
MeSH Terms: conditions — Opioid-Related Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Patients will come to the lab on 3 consecutive weekly visits. On the first, they go through the consent process and if signed, will have a clinical interview and ROS then be given baseline measures and then treated with transcranial photobiomodulation, following which they will undergo post-treatment measures. The treatment the first week will be randomized to active or sham and the second week they will receive the opposite treatment. The third week will be a follow-up of the second treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: One experimenter will act as the blinder and treater. Only he will know whether the patient receives the active or sham treatment and only he will prepare and provide the treatment. The patient and outcomes assessors will be blind to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active (Active Comparator): Patients will receive the active treatment.
  Interventions: Device: unilateral transcranial photobiomodulation, near infrared mode
- Sham (Sham Comparator): Patients will receive the sham treatment (the identical LED covered by aluminum foil).
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: unilateral transcranial photobiomodulation, near infrared mode — The investigators are applying a supra luminous LED at 810 nm and 250 mW/cm2 to the forehead of the participant at F3 and F4.
  Arms: Active
Device: Sham treatment — The sham treatment is identical to the active treatment except that the sham treatment has a piece of aluminum foil covering the led so that the participant will experience warmth but receive no photons.
  Arms: Sham

SUMMARY:
The investigators wish to test the hypothesis that transcranial photobiomodulation (tPBM) (i.e., 4-minutes of 810nm near-infrared light at 250 mW/cm2 by LED to the forehead at F3 or F4 versus an indistinguishable placebo treatment) can safely reduce opioid craving in individuals with opioid dependence in a within-patient study.

DETAILED DESCRIPTION:
Opioid use disorders (OUD) are an epidemic causing catastrophic consequences to individuals, families, and society despite treatments including psychotherapy, substitution therapy or receptor blockers, and psychoeducation. The investigators have developed a novel treatment that combines transcranial photobiomodulation (t-PBM) and Schiffer's Dual Brain Psychology (DBP)

The investigators will use a randomized, double-blind, placebo-controlled protocol in which 22 patients with significant opioid cravings and a history of recent or current OUD attended three one-hour weekly sessions. After baseline measures of opioid craving, and other psychometrics, subjects will receive two unilateral t-PBM applications (810 nm CW LED, 250 mW/cm2, 60 J/cm2, 4 min) or a sham (foil-covered LED) at F3 or F4. Prior to any treatment, the investigators will use 2 tests to determine which hemisphere is more associated with a negative outlook and cravings and will treat that side before the more positive hemisphere. The primary outcome measure will be an opioid craving scale (OCS). plus weekly Hamilton Depression (HDRS) and Anxiety (HARS) Rating Scales prior to treatments. Patients will be closely monitored for any possible adverse side-effects from the treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients complain of opioid cravings
* between the ages of 18 and 65.
* meet criteria for a history of opioid dependence by DSM V.

Exclusion Criteria:

* a past history of a psychotic disorder (including schizophrenia or schizoaffective disorder)
* a history of violent behavior
* a history of a past suicide attempt
* a history of current suicidal ideation
* a history of a neurological condition (e.g. epilepsy, traumatic brain injury, stroke), pregnancy,
* any current acute or chronic medical condition that might confound the study.
* Any patient judged by an investigator to have an impaired decision-making capacity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Opioid Craving Scale, OCS | immediately before and after treatments and one week later
  A published scale that consists of 3 questions, each rated by the patient from 0 to 9. with 9 indicating severe cravings.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale, HDRS | Before each treatment and 1 week later
  Standard depression rating scale; 0 to 53, a low score is less depressed. 0 to 7 is no depression.
Hamilton Anxiety Rating Scale, HARS | Before each treatment and 1 week later
  A standard anxiety rating scale; 0 to 56, a lower score suggests less anxiety
The Positive and Negative Affect Scale, PANAS | Before each treatment and 1 week later
  Patient rated positive and negative affects from 1 to 5. Five indicates extreme positive or negative affect. Scores for Positive and Negative Affects range from 0 to 25. A higher positive affect score and a lower negative affect score are better.

CONTACTS AND LOCATIONS:
Overall Officials: Fredric Schiffer, Principal Investigator — MindLight, LLC
Locations (1):
- MindLight, LLC, Newton Highlands, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
No personal identifying information of the patients will ever be released, but data for patient numbers will be.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available publication of the study and will be available online if the study is published.

REFERENCES:
- See also: published paper describing the study — https://www.frontiersin.org/articles/10.3389/fpsyt.2020.00827/full